Cover Page
Type of Document: Study Protocol
Official Title of the study: Integrating Alcohol Myopia and Objectification to Understand Sexual
Assault

NCT number: NCT03956238 Date of document: 2-28-20

Study 1: Sexual Objectification and Alcohol-Involved Sexual Aggression (Aim 1) Participants and procedures. Study 1 will utilize a mixed model experimental design with intoxication (alcohol, placebo control) as the between-participants factor and eye tracking and implicit association tests used to assess objectification as within-participants factors. We expect the behavioral manifestations of myopia—impaired attention and sexual objectification— will emerge in the intoxication condition compared to the placebo control condition. Specifically, community men (n = 150) will come to the lab for a study on "alcohol and perceptions" and be randomized to consume a moderate-dose alcohol or placebo drink, after which they will complete the attention, objectification, and sexual aggression measures.

**Alcohol administration.** Standard alcohol administration procedures used by the PIs in prior studies (e.g., Watkins, DiLillo, & Maldonado, 2015) will be employed. Men in the alcohol condition will be administered a dose of .90 g(amount of alcohol)/kg(men's weight) of 95% alcohol U.S. Pharmacopoeia (USP) mixed at a 1:5 ratio with a mixer to achieve a target BAC of at least .08%. Four milliliters of alcohol will be added to the mixer and alcohol will be sprayed on the rim of placebo beverages. All participants will have up to 30 minutes for beverage consumption. For participants in the alcohol condition this will be followed by a 20-minute absorption period. Because the effectiveness of alcohol placebo manipulations tends to diminish starting at about 30 minutes after beverage consumption (Bradlyn & Young, 1983), participants in the placebo condition will have a shorter, 10-minute absorption period.

**Attentional capacity.** Reduced attentional capacity associated with alcohol myopia will be assessed with the 5-item Mindful Attention Awareness Scale-State version (MAAS-S, Brown & Ryan, 2003). The MAAS-S assesses mindful attention (or lack thereof, I was doing something automatically without being aware of what I was doing) in the present moment or recent past (0 = not at all, 3 = somewhat, 6 = very much). The MAAS has high internal reliability ( $\alpha$  = .92) and demonstrates construct validity through associations with decreased attentional capacity on the operation span task (Black, Semple, Pokhrel, & Grenard, 2011). Within our myopia framework, we expect intoxication will cause self-reported difficulty paying attention.

**Objectification.** Given the central role of objectification in this model, this construct will be assessed multi-modally, using behavioral, implicit, and self-report measures (to capture explicit as well as covert attitudes of which people may be relatively unaware or fail to report due to social desirability). Behavioral assessment will occur with the Eye-Tracking Objectification Task (Gervais et al., 2013), to assess objectifying gazes. A portable eye-tracking system is used to measure participants' gazes toward a woman. Specifically, men are told that they are completing a study of media preferences with another participant, an attractive woman wearing revealing clothing. In a series of scripted interactions with the woman, the participant learns that the woman dislikes media with sexual content (which serves as the foundation for the sexual aggression measure, see below). Of interest here will be participants' gazes toward the woman's face and body (and sexual body parts in particular, e.g., breasts). Within the context of the myopia framework, attention to the woman's body represents a provoking cue, whereas attention to the woman's face represents an inhibiting cue. Intoxication is expected to increase objectifying gazes.

Participants will also complete the Female Object Brief-Implicit Association Task (female object B-IAT, Rudman & Mescher, 2012), which provides a measure of implicit objectification of women (associating women more with objects vs. humans). Implicit associations are assessed by presenting words from different categories (e.g., women, objects, humans) and asking people to press the same response key for two categories of words (e.g., pressing "e" whenever

a "woman" word [e.g., female] or an "object" word [e.g., tool] appears on the screen vs. pressing "e" whenever a "woman" word or a "human" word [e.g., person] appears). Making a response is easier (and thus faster) when closely related constructs share the same response key. Therefore, quicker response times when woman and object (vs. human) words are paired represents more implicit objectification. We expect intoxication to cause faster reaction times when women and object words are paired and slower reaction times for pairings of women and human words.

The Other-Objectification Questionnaire (modified from Grabe, Routlege, Cook, Andersen, & Arndt, 2005; Curran, 2005), which assesses the frequency (6=very frequently, 1=never) with which the male participant objectified the female confederate (e.g., I focused more on her body than our conversation). Scores are averaged with higher scores representing more objectification of women. We expect intoxication to cause more weight to be placed on women's objectifying compared to human attributes in men's evaluations.

Sexual aggression. To assess sexual aggression, participants will complete the Laboratory Analogue of Sexual Aggression (Parrott et al., 2012) based on Hall, Hirschman, and Olivier (1994). Following the ostensible interaction in which the participant learns that the female participant dislikes media with sexual content, men then select one clip—containing either a man and a woman having sexual intercourse or a similar clip without sexual content—for the woman to watch based on still shots and synopses. Choosing the sexual (vs. non-sexual) clip represents sexual aggression. Although perpetrators may justify their choices (e.g., reasoning that the woman may not like sexual content in general, but that she would like this sexual content in particular), such responses fall under the CDC definition of sexual violence (i.e., subjecting a woman to an unwanted sexual experience). Validity of the paradigm is supported by expected positive associations between selection of the sex video and self-reported history of sexual aggression perpetration, adversarial heterosexual beliefs, hostility toward women, and hostile sexism (Parrott et al., 2012). We expect intoxication to cause more sexual aggression.

Study 2: Self-Objectification and Alcohol-Involved Sexual Victimization (Aim 2) Participants and procedures. Study 2 will use a mixed model experimental design with intoxication (alcohol, placebo control) and objectification (objectifying gazes, eye contact control) as between-participant factors and implicit association tests used to assess self-objectification as within-participant factors. The effects of intoxication and objectification on impaired attentional capacity, self-objectification, and victimization risk perceptions in a representative sample of 210 community women will be assessed. Participants will come to the lab for a study of "alcohol and perceptions," providing a cover story for the alcohol and objectification manipulations and attention, self-objectification, and victimization risk measures.

**Alcohol administration.** Randomization to the alcohol conditions (alcohol, placebo control) will be identical to those in Study 1 with two exceptions. Because of gender differences in body fat composition, women will be given a dose of .85 g(amount of alcohol)/kg(men's weight) of alcohol in the alcohol condition (Giancola et al., 2002).

**Objectification.** To parallel men's objectification behaviors, we will use the objectifying gaze lab paradigm developed and validated by PI Gervais (Gervais, et al., 2011, 2016; Kimble et al., 2016; Wiener, Gervais et al., 2013). During a getting acquainted interview, a male confederate (ostensibly another participant) will be randomized to either: (a) engage in objectifying gazes directed at women's breasts lasting 2-3 seconds at several points, or (b) maintain eye contact

with the participant. The confederates undergo rigorous training to deliver the gazes consistently over time and across participants in a natural manner, and perceptions of the confederate (e.g., attractiveness) are collected and controlled for in analyses.

**Attentional capacity.** As in Study 1, the 5-item self-report Mindful Attention Awareness Scale-State (MAAS-S, Brown & Ryan, 2003) will be used to assess impaired attentional capacity. We expect that intoxication will cause more impaired attention capacity on the MAAS-S.

**Self-objectification**. Similar to sexual objectification for men, self-objectification will be assessed in three complementary ways. A portable eye-tracking system will be used to measure participants' gazes toward their own bodies. Specifically, a mirror will be present in the room during the objectifying gaze lab paradigm. While women are interacting with the male confederate and shortly thereafter, women's gazes toward their own faces and bodies will be assessed with a portable eye tracker. Intoxication and objectification from the male confederate is expected to increase self-objectifying gazes.

Participants will also complete the 10-item Self-Objectification Questionnaire (SOQ; Noll & Fredrickson, 1998). Participants rank order objectifying appearance (e.g., sex appeal, appearance) and non-objectifying, human (e.g., health, stamina) attributes in order of importance (0 = least, 9 = most) to their self-concept. Rankings on non-observable, internal attributes are subtracted from observable, objectifying attributes with higher scores representing more self-objectification. The SOQ is a widely used measure of self-objectification with demonstrated validity (Calogero, 2011). We expect that intoxication and objectification will cause more self-objectification on the SOQ.

Similar to Study 1, participants will also complete the Self-Object Brief-Implicit Association Task (self-object B-IAT; Morris, Goldenberg, & Heflick, 2014), which provides a measure of implicit self-objectification (associating the self more with objects than humans). With the Self-Object B-IAT, "self" (instead of "woman") words (e.g., me, self) are paired with object words or human words. Faster response times when self and object (vs. human) words share a response key represents more implicit self-objectification. We expect intoxication and objectification to cause more self-objectification on the B-IAT.

Risk for sexual victimization. Due to the ethical proscriptions against replicating sexual victimization in the lab, we will assess risk for victimization using the Risk Perception Survey (RPS; Messman-Moore & Brown, 2006). The RPS consists of vignettes depicting forced sexual intercourse. The vignettes include clear (sexual comments, male persistence) and ambiguous (alcohol consumption, physical isolation) risk factors. They contain chronological statements that become progressively riskier as the man increases his coercion. Respondents imagine themselves interacting with the man and the RPS yields a "leave" variable, which reflects the point at which the participant indicates she would leave. We expect impaired risk perception as indicated by higher "leave" values when women are intoxicated and objectified.

## Objectification and Alcohol-Involved Sexual Assault: Critical Moderators (Aim 3).

To address Aim 3, participants in Study 1 and Study 2 will complete measures of key moderators online prior to coming to the lab. In Study 1 men will complete the 10-item Sexual Experiences Survey-Short Form Perpetration (SES-SFP; Koss et al., 2007). The SES-SFP assesses the frequency (0 to 3+) of unwanted sexual contact, coercion, attempted rape, and rape. Men will also complete the 10-item Other-Objectification Questionnaire (OOQ) in which

they will rank order the importance of 10 objectifying attributes (e.g., sex appeal) and humanizing, internal attributes to assess overall objectification of women (Noll & Fredrickson, 1998; Grabe et al., 2005; e.g., relative importance of sex appeal vs. well-being, internal states, attributes in women). The ranking for the human attributes is subtracted from the ranking of the objectifying attributes with higher numbers indicating greater objectification of women.

Women in Study 2 will complete the 10-item Self-Objectification Questionnaire (SOQ; Noll & Fredrickson, 1998) that uses the same items, response format, and scoring procedure as the OOQ, except people are asked to rank the objectifying and human attributes in themselves to assess self-objectification. Sexual victimization will be assessed with the 10-item Sexual Experiences Survey-Short Form Victimization; SES-SFV; Koss et al., 2007), which assesses the frequency of unwanted sexual advances using the same format as the SES-SFP, but with items worded for victimization rather than perpetration.

Both men and women will complete the 18-item Sex-Related Alcohol Expectancies Scale (SRAES, Dermen & Cooper, 1994), that assesses the degree to which people associate alcohol consumption with sexual disinhibition and risk (e.g., I have sex with people whom I wouldn't have sex with if I were sober) on 6-point scales (1 = strongly disagree, 6 = strongly agree). The SRAES is psychometrically sound including adequate internal consistency reliability ( $\alpha$  = .70 - .83) and is correlated with alcohol use and sexual risk-taking (Dermen & Cooper, 1994). Men and women will also complete the 19-item Rape Myth Acceptance Scale (RMAS, Burt, 1980), which assesses people's support of rape myths (e.g., Any healthy woman can successfully resist a rapist if she really wants to) on 7-point scales (1 = strongly disagree, 7 = strongly agree).

We expect the predicted effects to be most pronounced for men high on objectification and with a history of sexual assault perpetration (Study 1) and for women high on self-objectification and with a history of sexual assault victimization (Study 2). We also expect these effects to be more exaggerated for men (Study 1) and women (Study 2) high in sex-related alcohol expectancies and rape myth acceptance.